CLINICAL TRIAL: NCT06334081
Title: Clinical Outcomes of Two Different Surgical Drilling Protocols of Immediate Loaded Dental Implant in Posterior Maxilla
Brief Title: Different Surgical Drilling Protocols in Posterior Maxilla
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Elsheikh, assistant professor of oral and maxillofacial surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A02040230S
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Missing Teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A dental implant placement by undersized drilling technique. (Experimental): 8 dental implants placed in the healed alveolar posterior maxillary ridge using undersized drilling technique
  Interventions: Procedure: undersized drilling technique
- Group B dental implant placement by single drilling technique (Experimental): 8 dental implants placed in the healed alveolar posterior maxillary ridge using singledrilling technique
  Interventions: Procedure: single drilling technique

INTERVENTIONS:
Procedure: undersized drilling technique — In group A The implant site preparation was made according to the protocol of the manufacturer except that the final drill was omitted. The drilling was done using a low speed reduction, high torque with coolant contra-angle hand piece with surgical motor unit. Speed of drilling was 800-1200 rpm.
  Arms: Group A dental implant placement by undersized drilling technique.
Procedure: single drilling technique — In group B The implant bed was prepared using the new specially designed drills. First, the use of the guide drill of length 3.5mm with speed of 800 rpm and torque of 35 nm, then the use of the one drill of the same diameter of the selected implant size to the full length of the osteotomy site.
  Arms: Group B dental implant placement by single drilling technique

SUMMARY:
Sixteen dental implants inserted in sixteen patients who were selected from the outpatient clinic of the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University, for the rehabilitation of missed single maxillary posterior tooth by an immediately loaded dental implants

DETAILED DESCRIPTION:
16 dental implants were inserted in 16 patients were divided into two groups: Group A: 8 dental implants were inserted using undersized drilling technique and Group B: 8 dental implants were inserted using single drilling technique. then the dental implants were assessed for 6 months regarding

Clinical Evalution: regarding these parameters after immediately dental implants loading,3 months and 6 months.

implant stability, implant probing depth, bleeding index.

Radiographic evaluation: immediately after implant loading and 6 months after loading regarding bone density and marginal bone loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients with missed one or more posterior maxillary tooth.
* Be older than 18 years and of residual bone height more than10 mm.
* Patients with good oral hygiene and willing to participate in the follow-up sessions.
* Patients with adequate mesio-distal width and inter-arch space.
* Patients without any para-functional habits such as clenching and bruxism.

Exclusion Criteria:

* Patients whose proposed surgical site had any pathological lesion or root tips.
* Drug or alcohol abuse.
* Patients with uncontrolled systemic diseases.
* Pregnant patients.
* Tobacco use more than fourteen cigarettes daily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
bone density measurement | 6 month
  cbct will be done to evaluate difference in bone density
marginal bone loss | 6 month
  cbct will be done to evaluate marginal bone loss

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Elsheikh, Al Mansurah, Egypt